CLINICAL TRIAL: NCT05873205
Title: Open-Label, Phase II Trial of Isatuximab for Patients With Refractory Immune Cytopenias After Allogeneic Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-119
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Blood Cancer; Refractory Immune Cytopenias
Keywords: Refractory Immune Cytopenias; Blood Cancer; Isatuximab; Allogeneic Hematopoietic Cell Transplantation; 23-119; Memorial Sloan Kettering
MeSH Terms: conditions — Hematologic Neoplasms | interventions — isatuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants with Refractory Immune Cytopenias (Experimental): Participants will be adults who develop Immune Cytopenias/ICs after Allogeneic Hematopoietic Cell Transplantation/allo-HCT and who did not respond to initial immunosuppressive therapy.
  Interventions: Biological: Isatuximab

INTERVENTIONS:
Biological: Isatuximab — All participants enrolled on the study will receive isatuximab intravenously as a single agent

SUMMARY:
The purpose of this study is to find out whether isatuximab is an effective treatment for people who developed immune cytopenias/ICs after allogeneic hematopoietic cell transplant/allo-HCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (There are no dosing/AE data for isatuximab in children).
* Disease for which patient underwent an allo-HCT is in documented remission.
* Patients must have previously had documented primary neutrophil and platelet engraftment, defined as:

  * Neutrophil engraftment: the first of 3 successive days with an absolute neutrophil count of ≥500/μL after post-transplantation nadir.
  * Platelet engraftment: the first of 3 consecutive days with a platelet count of 20,000/μL or higher in the absence of platelet transfusion for 7 consecutive days.
* Patients must be at least 45 days post allogeneic HCT to enroll.
* Patients must be diagnosed with IC(s) based on the following criteria:

  o For AIHA: Positive (abnormal) DAT test and decreasing hemoglobin of ≥2 g/dL from a stable baseline (i.e., from the patients typical hemoglobin value prior to AIHA) and at least grade 2 (i.e., hemoglobin <10 g/dL) due to evidence of hemolytic anemia with ≥2 of the following tests: increased reticulocyte count (>ULN), increased lactate dehydrogenase (LDH) (>ULN), decreased haptoglobin (<LLN), increased unconjugated bilirubin (>ULN).
* DAT negative AIHA may be included providing exclusion of alternative etiology of hemolytic anemia.

  * For ITP: decreasing thrombocytopenia from baseline (i.e., from the patients typical platelet count prior to ITP) and platelet count ≤30 K/µL or requiring platelet transfusions in the absence of other causes of thrombocytopenia (including drug-induced thrombocytopenia), and with normal or increased bone marrow megakaryocytes.
  * For PRCA: severe anemia (hemoglobin <8 g/dL without transfusions) with reticulocytopenia (reticulocyte percentage <1% and/or absolute reticulocyte count <10,000/µL) after exclusion of obvious causes of anemia.
  * Patients with concomitant ICs can be enrolled on the study.
* Patient must have responded incompletely to their previous treatment, defined as:

  * Corticosteroid refractoriness: defined as a clear progression or minimal responsiveness of IC(s) after ≥7 days of treatment with prednisone equivalent of ≥1 mg/kg/day.
  * Corticosteroid dependence: defined as dependence on prednisone equivalent of ≥0.5 mg/kg/day to maintain hemoglobin level ≥2 g/dL nadir level (for AIHA and/or PRCA), and/or platelet count ≥30 x 109/L or ≥2-fold increase from nadir level (for ITP).
  * Refractory IC(s) after ≥2 treatment lines including corticosteroids (≥0.5 mg/kg/day prednisone equivalent), IVIG (400 mg/kg/day for 2 to 5 days), and/or rituximab, etc.

    * For rituximab treated patients, refractoriness will be defined as no or minimal response within 2 weeks of completing ≥4 doses of rituximab.
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L.

  o Growth factors, including granulocyte colony stimulating factors and erythropoietin are allowed, but should be administered at a stable dose.
* No active hepatitis viral infection or on active treatment for hepatitis infection.
* Female patients of childbearing potential are eligible if the patient has had a negative serum or urine pregnancy test within 10-14 days prior to starting isatuximab therapy.

They must also agree to avoid pregnancy by using an adequate method of contraception (2 barrier method or 1 barrier method with a spermicide or intrauterine device) for 2 weeks prior to screening, during and 5 months after the last dose of trial medication. Adequate methods of contraception are provided as examples. Other acceptable and effective methods of birth control are also permitted (e.g., abstinence).

* Male patients must agree to not donate sperm while on the study and for at least 5 months after the last dose of study drug. They must agree to use contraception during the intervention period and for at least 5 months after the last dose of isatuximab treatment.
* Subjects must be able to give informed consent.

Exclusion Criteria:

* Presence of relapse/progression of malignant disease for which the patient underwent allo-HCT
* Patients with anemia and/or thrombocytopenia related to transplant-associated thrombotic microangiopathy.
* Patients with active GVHD requiring therapy may be eligible if the GVHD is responsive to treatment (< grade 4 in severity), and after agreement between the sponsor and principal investigator.
* Organ insufficiency based on above criteria.
* Pregnancy or unwillingness to agree to birth control as noted above.
* Known to be HIV+ or to have active hepatitis A, B, or C infection (i.e., with viremia).

Of note:

* Patients can be eligible if anti-HBc seropositive (with or without positive anti-HBs), but HBsAg and HBV DNA are negative.
* Patients with antiviral therapy for HCV started before initiation of treatment and positive Hep C antibodies are eligible. The antiviral therapy for Hep C should continue throughout the treatment period until seroconversion. Patients with positive anti-Hep C and undetectable Hep C RNA without antitviral therapy for Hep C are eligible.

  * Any clinically significant, uncontrolled medical condition(s), including infection(s) that, in the Investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
  * Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose, prior anti-CD38 moAb such as daratumumab, or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
  * Received any investigational drug within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer. In case of very aggressive disease (e.g., acute leukemia) delay could be shortened after agreement between sponsor and principal investigator, in absence of residual toxicities from previous therapy.
* Patients on post-HCT maintenance therapy to reduce the risk of relapse (for patients with hematologic malignancies) or GVHD (e.g., FLT3 inhibitors, etc.) may be eligible after agreement between the sponsor and principal investigator.

  * Contraindication to any concomitant medication, including pre-medications or hydration given prior to therapy
  * Participants who are unable to consent to the study or comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 4 years
  To estimate the overall response rate (ORR; complete response [CR] + response)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scorder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org